CLINICAL TRIAL: NCT01652898
Title: A Single Centre Prospective, Randomized, Double Blind, Crossover, Three-treatment Periods PK, PD, Safety and Tolerability Study to Compare Bolus Administration of AOP LDLA202, ONO LDL50 and Esmolol in Healthy Volunteers After a Pilot Phase of AOP LDLA202 Safety and Local Tolerability Assessment.
Brief Title: A Pharmacokinetic, Pharmacodynamic, Safety Study With AOP LDLA202, ONO LDL50 and Esmolol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOP LDLA202.101
Record Dates: First submitted 2012-07-19; First posted 2012-07-30 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: PK
MeSH Terms: interventions — esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Esmolol hydrochloride (Active Comparator): Esmolol hydrochloride administered as intravenous bolus injection at low (0,5mg/kg), medium (1mg/kg) and high dose (1,5mg/kg) in 15/30/45 seconds once per subject
  Interventions: Drug: Esmolol hydrochloride
- ONO LDL50 (Active Comparator): ONO LDL50 administered as intravenous bolus injection at low (0,1mg/kg), medium (0,2mg/kg) and high dose (0,3mg/kg) in 15/30/45 seconds once per subject
  Interventions: Drug: ONO LDL50
- AOP LDLA202 (Experimental): AOP LDLA202 administered as intravenous bolus injection at low (0,1mg/kg), medium (0,2mg/kg) and high dose (0,3mg/kg) in 15/30/45 seconds once per subject
  Interventions: Drug: LDLA202

INTERVENTIONS:
Drug: LDLA202 — Comparison of 3 different doses LDLA202, 40 PK samples, 40 BP and ECG measurement time points, 23 local tolerability measurement time points
  Arms: AOP LDLA202
Drug: ONO LDL50 — Comparison of 3 different doses ONO LDL50, 40 PK samples, 40 BP and ECG measurement time points, 23 local tolerability measurement time points
  Arms: ONO LDL50
Drug: Esmolol hydrochloride — Comparison of 3 different doses Esmolol, 40 PK samples, 40 BP and ECG measurement time points, 23 local tolerability measurement time points
  Arms: Esmolol hydrochloride

SUMMARY:
The study consists of a Pilot Phase (to assess safety and the local tolerability of highest AOP LDLA202 dose versus placebo) and a Main Treatment Phase (to compare PK, PD and safety and tolerability of AOP LDLA202, ONO LDL50 and esmolol bolus administrations by measurement of blood concentrations of landiolol, esmolol and their metabolites, and by monitoring ECG, blood pressure and adverse events).

DETAILED DESCRIPTION:
A single centre prospective, randomized, double blind study consisting of a local safety Pilot Phase and a triple-cross-over Main Study Phase.

In the pilot phase, 3 subjects will be administered a bolus with AOP LDLA202 vs. placebo (0.9% saline) simultaneously (same vein on the other body side). Following treatment of the first subject per cohort and assuming no safety concerns arise, second and third subjects will be treated in safety intervals of at least 3 hours between doses in individual subjects. On Day 3 after dosing a safety follow-up assessment will be done and all adverse events will be reported to the sponsor's medical monitor. Assuming no safety concerns arise, the sponsor's medical monitor will give green light for conduct of the Main Treatment Phase in writing.

In the main phase, 12 subjects will be treated with AOP LDLA202, ONO LDL50 and esmolol. Three doses per subject and day (=treatment period), all administered via big superficial veins, are planned with at least 1 hour observation period after each bolus injection. Each subject, if confirmed eligible, will complete three treatment periods in total in the main phase of the study.

ECG, blood pressure, local tolerability and adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Male and female human subjects, age 18-45 years, Caucasians
* Body weight of at least 50 kg, maximum of 90 kg. Body-mass index 18.5 to 30.0 kg/m2.
* Subjects without clinically relevant abnormalities as determined by baseline medical history, physical examination, blood pressure, heart rate and ear temperature at screening.
* Subjects without clinically relevant abnormalities as determined by blood count, coagulation tests, biochemistry, infectious disease screening, urinalysis, ECG, and 2D Echo at screening.
* Subject is willing and able to undergo procedures required by this protocol and gave written informed consent.
* Agreeing to not using any prescription and over the counter medications
* No history or presence of alcoholism or drug abuse

Exclusion Criteria:

* Subjects with history or presence of clinically relevant cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, hematological, gastrointestinal, endocrine, immunological, psychiatric or skin diseases.
* Subjects with bradycardia (heart rate below 50 bpm), tachycardia (heart rate above 100 bpm), hypotension (systolic blood pressure below 100 mmHg, and/or diastolic blood pressure below 70 mm Hg) at screening, history of clinically relevant arrhythmias.
* Subjects with clinically relevant cardiac supraventricular or ventricular arrhythmias.
* Subjects with atrioventricular block of grade II and III, sick sinus syndrome, sinoatrial block or congestive heart failure.
* Participation in a clinical drug study or bioequivalence study 60 days prior to present study.
* History of malignancy or other serious diseases.
* Any contraindication to blood sampling.
* History of i.v. drug abuse.
* Subjects with positive HIV tests, HBsAg or Hepatitis C tests or other acute, subacute or chronic infectious disease.
* Known history of hypersensitivity to any IMP.
* Refusal to abstain from smoking or consumption of tobacco products 48 hours before drug administration and during the study period.
* Refusal to abstain from alcohol, caffeine, or other xanthines, or grapefruit containing food or drinks for 72 hours before drug administration and during the study period.
* Refusal to abstain from strenuous activities for 7 days before screening and end-of-study examinations, before and during each study period.
* Subjects with anomalies of the venous and arterial vessels of the forearms or systemic vascular diseases.
* Pregnancy and/or breast-feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
PK as measured by Cmax, Tmax, AUC, residual area, T1/2, CL and V | 7 hours
Local tolerability as measured by signs and symptoms of inflammation judged by the clinical investigator on a 6-symptom, 4-point venous score. | 7 hours
Safety as measured by Adverse events, clinical chemistry, hematology, urinalysis, physical examination, ECG (HR, PQ (PR), QRS, QT and QTc) and BP in mmHg. | 7 hours

SECONDARY OUTCOMES:
PD as measured by BP in mmHg and ECG parameters (HR, PQ, QRS, QT and QTc) | 7 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Ulc, Dr. med., Principal Investigator — Cepha s.r.o
Locations (1):
- Cepha s.r.o, Pilsen, Czechia

REFERENCES:
- [Derived] Krumpl G, Ulc I, Trebs M, Kadlecova P, Hodisch J. Bolus application of landiolol and esmolol: comparison of the pharmacokinetic and pharmacodynamic profiles in a healthy Caucasian group. Eur J Clin Pharmacol. 2017 Apr;73(4):417-428. doi: 10.1007/s00228-016-2176-0. Epub 2017 Jan 13. PMID 28091703
- See also: Sponsor — http://www.aoporphan.com/